CLINICAL TRIAL: NCT03791697
Title: Preferred Method of Postoperative Follow Up After Pelvic Reconstructive Surgery. (Phone Call Versus Clinic Visit): A Non-Inferiority Randomized Clinical Trial
Brief Title: Telehealth Postop Follow up RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jackson, Elisha (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Principal Investigator, Elisha Jackson, Physician-Fellow, Jackson, Elisha
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Telehealth Study
Record Dates: First submitted 2018-12-30; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Patient Satisfaction
Keywords: Postoperative patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to Arm1 or Arm2 (Telephone follow up or clinic follow up). Permuted block randomization with randomly varying block sizes will be used. Generation of allocation sequences will be performed using a random-number table.
  The allocation sequence will be generated by our statistician who is neither responsible for patient recruitment or outcome assessment. Sequentially numbered opaque sealed envelopes will be used for concealment of treatment allocation.
  It is not possible to mask clinical staff or participants, as they will be aware of the follow-up care that is being delivered over the telephone or in clinic. As such this is not a blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Group (Active Comparator): The patient randomized into the telephone follow up group, will be contacted, at the pre-scheduled date and time, by the urogynecology clinic nurse. The nurse will utilize a scripted series of postoperative questions, which are consistent with questions asked during our standard postoperative clinic visits.
  Vital signs and physical examination will be deferred for the patients in the telephone follow up group.
  Any patient responses that are not consistent with a usual postoperative course will be escalated to an in person visit. However, these patients will remain in the group, to which they were originally randomized, for research analysis purposes.
  Interventions: Other: Telehealth 2 week postoperative visit
- In Person Clinic Visit Group (No Intervention): For the patient randomized into the clinic group, the clinic visit will entail questions about common postoperative complications (including fever, nausea/vomiting, pain, urinary symptoms, constipation, etc.). As per usual, vital signs and a focused physical examination will be completed at the clinic visit. All clinic visits will be performed by an FPRMS fellow and/or attending physician

INTERVENTIONS:
Other: Telehealth 2 week postoperative visit — The patient randomized into the telephone follow up group, will be contacted, at the pre-scheduled date and time, by the urogynecology clinic nurse. The nurse will utilize a scripted series of postoperative questions, which are consistent with questions asked during our standard postoperative clinic visits.
  Vital signs and physical examination will be deferred for the patients in the telephone follow up group.
  Any patient responses that are not consistent with a usual postoperative course will be escalated to an in person visit. However, these patients will remain in the group, to which they were originally randomized, for research analysis purposes. (Intent to treat)
  Arms: Telephone Group

SUMMARY:
A randomized controlled trial that will evaluate whether telephone two-week postoperative follow up visits are an acceptable and safe alternative to traditional face-to-face-clinic two-week postoperative visits.

DETAILED DESCRIPTION:
This is a two group, parallel randomized non-inferiority clinical trial at one institution evaluating telephone postoperative visits as non-inferior in patient satisfaction, patient preference, and patient safety, when compared with clinic postoperative visits. This protocol was written in accordance with CONSORT (Consolidated Standards of Reporting Trials) guidelines 2011.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 desiring surgical management of prolapse or incontinence
* English speaking
* Willing and able to provide written and informed consent without assistance from medical surrogate or interpreter
* Immediate access to telephone services (landline, mobile phone, office phone)

Exclusion Criteria:

* Women <18
* Non-English speaking
* Unwilling and unable to provide written and informed consent without assistance from surrogate or interpreter
* Hearing impairment
* No access to telephone services (landline, mobile phone, office phone)
* Grade 3 complication- a complication requiring surgical, endoscopic, or radiological intervention. [3]
* Patient who did not attend any postoperative follow up visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction (questionnaire) | Survey will be provided at the six-week follow up visit.
  Comparison of patient satisfaction as determined by completion of a non-validated, treatment non-specific satisfaction questionnaire between the two groups.

SECONDARY OUTCOMES:
Patient safety (adverse events) | Postoperative period up to 6 weeks
  • Comparison of adverse events and Emergency Department (ED) visits between the two groups. Will be determined by reviewing the patient's record to identify adverse events as defined below
Time Spent (post op telephone follow up compared to clinic follow up [minutes]) | Calculated from time spent at the two week follow up visit
  • Actual time spent on phone call during postoperative telephone follow up compared to time spent in clinic follow up measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Elisha J Jackson, MD, Principal Investigator — University of South Florida Morsani School of Medicine
Locations (1):
- University of Florida Health, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT03791697/Prot_SAP_000.pdf